CLINICAL TRIAL: NCT03817294
Title: Personalised Exercise Training in COPD - Exploring the Interaction Between Exercise Physiology, Exercise Perception and Training Progression
Brief Title: Personalised Exercise Training in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Tom Ward, Clinical PhD student, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS 243125
Record Dates: First submitted 2018-10-02; First posted 2019-01-25 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This a pilot/feasibility study, aiming to characterise exercise limitation at baseline and then conducting an abridged RCT with 4 training arms. The main outcomes are related to training progression and perception
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Eccentric cycling (Active Comparator)
  Interventions: Other: Comparison of exercise training modalities
- Concentric cycling (Active Comparator)
  Interventions: Other: Comparison of exercise training modalities
- Single leg cycling (Active Comparator)
  Interventions: Other: Comparison of exercise training modalities
- Lower limb resistance training (Active Comparator)
  Interventions: Other: Comparison of exercise training modalities

INTERVENTIONS:
Other: Comparison of exercise training modalities — As above

SUMMARY:
Exercise training as part of Pulmonary Rehabilitation (PR) has been shown conclusively to improve breathlessness,quality of life and exercise capacity for people with COPD. However generally PR is delivered in a 'one size fits all' approach without considering different aspects of an individual's disease. It is hypothesised that a more personalised approach to PR may yield even better results. However to design a personalised programme of PR we need a better understanding of how different people with COPD respond to different possible exercise training modalities. This study will therefore comprehensively characterise a group of patients and then ask them to complete 3 weeks of exercise training in one of four modalities; conventional cycling, eccentric cycling, one-legged cycling and resistance training. The aim is not to prove which type of training is more effective but to develop an idea of which groups of patients would benefit from which type of training.

Baseline measures would be designed to fully understand how an individual responds to exercise and would therefore be comprised of a variety of endurance tests, strength tests, questionnaires, and measurements of lung capacity and body composition. This is to give as much information as possible to identify different responses to exercise.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a highly prevalent condition affecting an estimated 1.2 million people in the UK and is the second most common lung disease after asthma. COPD not only affect the lungs, but is a systemic disease with muscle dysfunction being a significant feature. Exercise, as part of a programme of pulmonary rehabilitation (PR), has been shown to improve exercise capacity and quality of life of patients with COPD. However, despite the effectiveness of PR at a population level, there remains room for improvement. The individual treatment response is heterogeneous with some patients failing to achieve clinically significant improvements, whilst others struggle to adhere to the exercise component or drop out altogether. Currently, whilst exercise intensities (the "dose") are individualised during PR, the character and content of PR is generally provided in a "one size fits all" manner. There is therefore scope to modify the content of PR to meet individual needs and underlying physiology thereby enhancing adherence and benefits.

Precision medicine, tailoring therapy to specific "treatable traits" of an individual's condition, holds the potential to maximise treatment effect whilst minimising adverse effects. The investigators propose the same principles of precision medicine can be used to improve the delivery of PR by identifying an individual's exercise response at enrolment to PR and using this information to personalise exercise training. There are a growing number of diverse, novel training modalities that have been shown to be feasible and potentially efficacious in COPD, offering opportunities for delivering a personalised training programme. A key step in the development of this personalised/precision approach in exercise medicine is the understanding and measurement of the individual exercise pathophysiology that predicts preferential benefits to a particular exercise training modality. However, the relationship between baseline exercise pathophysiology (and indeed other disease and demographic variables) and such a response is currently unknown.

Eccentric exercise, contraction of a muscle as it lengthens, and one-legged cycling are two options for diversifying PR. For a given muscle workload, eccentric exercise results in lower energy demand and oxygen consumption and therefore puts less strain on the cardiopulmonary system. Consequently, this type of exercise may be ideally suited for patients with lung disease, particularly for those who stop exercise due to ventilatory limitations. It may be more tolerable for patients as it causes less breathlessness, whilst allowing greater muscle specific work. Eccentric cycling involves use of a bike with an attached motor which drives the pedals in reverse. The subject must resist the rotation of the pedals to maintain a constant pedal speed, thereby performing eccentric work with their legs. Using eccentric exercise as a training modality had historically been avoided due to the fear of causing muscle damage. High intensity eccentric resistance exercise leads to delayed onset muscle soreness (DOMS) and has been used for many years as a model of inducing muscle damage. However over the last 30 years there have been an increasing number of studies showing comprehensively that if load is gradually increased, muscle damage and soreness is minimal and acceptable. In patient populations, because loads achieved are particularly low, the occurrence of significant muscle damage is even more infrequent and previous work, has demonstrated that eccentric cycling is well tolerated in patients with COPD.

Whole body exercise, such as walking or cycling, requires recruitment of a large muscle mass generating a high oxygen demand. However, there is a disparity between whole body maximal oxygen uptake and muscle maximum aerobic capacity, even in a healthy population, and consequently significant variation in the muscle training stimuli achieved. This is emphasised in patients with COPD with a ventilatory limit to exercise. By exercising a smaller muscle mass, this ventilatory limitation can be bypassed and the individual muscle can be worked at significantly higher intensity. One method to reduce the exercising muscle mass is one-legged cycling. Two randomised controlled trials have demonstrated a greater improvement in V̇O2peak following one-legged cycling compared with two legged cycling in patients with COPD. One-legged cycling has been demonstrated to be a feasible addition to a PR programme and well received by patients and physiotherapists.

This study aims to determine how disease, demographic and exercise physiological variables recorded at baseline relate to subsequent perception and progression of novel training modalities compared to conventional training. The investigators will perform a comprehensive assessment of physiological response to exercise at baseline in terms of exercise capacity, exercise limitation, muscle volume and strength, physical activity, frailty and muscle composition. Participants will then be randomly allocated to one of 4 training modalities; eccentric cycling, one-legged cycling, concentric (traditional 2-legged cycling), or lower limb resistance training.

This is a pilot/feasibility study with the broad aim of identifying potential subphenotypes of patients with COPD that might respond preferentially to particular modalities of training. This knowledge is crucial to the development of definitive clinical trials of such exercise medicine interventions that could be delivered in routine clinical practice. The specific aims are:

1. To characterise in detail the underlying pulmonary and systemic pathophysiological characteristics of patients with COPD who are disabled by exercise limitation.
2. To measure progression of training loads during each training intervention relative to baseline values.
3. To determine how baseline characteristics and pathophysiology relate to training progression and exercise experience.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 40 years or above
* Diagnosis of COPD
* FEV1/FVC <0.7 and FEV1 < 80% predicted
* Medical Research Council (MRC) dyspnoea scale ≥3
* Participant is willing and able to give informed consent for participation in the study.
* Stable dose of current regular medication for at least 4 weeks prior to study entry.
* Participant has clinically acceptable ECG at enrolment.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* English speaking

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Any major or uncontrolled comorbidity that would impair the participant's ability to exercise or would mean exercise was unsafe.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks
* Participation in pulmonary rehabilitation in the preceding 6 months
* Participation in another research study involving exercise training in the preceding 6 months
* Acute exacerbation in the preceding 4 weeks (would become eligible 4 weeks following recovery)
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Training Progression (Total work during training relative to baseline) | 3 weeks
  (Total load during training in kJ or kg depending on exercise modality)/(load performed at baseline). This will therefore be presented as a standardised proportion (%) with no unit of measurement. Load refers to the total force production during exercise. For 2 leg and 1 leg concentric cycling and eccentric cycling this refers power output of the ergometer - total energy produced. For resistance exercise this refers to total weight lifted during training (in kg), i.e. weight lifted multiplied by number of repetitions.
Training adherence | 3 weeks
  (percentage of training sessions attended)
Subjective exercise experience scale during each exercise modality | Week 2
  Validated 12 point questionnaire with each question scoring from 1 (not at all) to 7(very much so). 3 domains - fatigue (high score=high fatigue), positive well-being (high score=high positive well being) and psychological distress (high score=high distress). Each domain represents 4 questions and the score for each domain (from 4-28) will be presented. Completed during all 4 exercise modalities (eccentric cycling, resistance training, single leg cycling and concentric cycling) for each participant

SECONDARY OUTCOMES:
Experience of different exercise modalities - Qualitative questionnaire | 3 weeks
  Structured questionnaire tailored to this study requiring short answers. Exploring preference and experience of each training modality. Note: This is not a scale questionnaire, but a short answer questionnaire with results presented as 'themes'
Exercise capacity - peak V̇O2 during a maximal incremental 2 leg cycle test | Baseline
  ml.min-1
Exercise capacity - peak V̇O2 during a maximal incremental 1 leg cycle test | Baseline
  ml.min-1
Inspiratory capacity during maximal 2 leg cycling | Baseline
  change from baseline (ml)
Functional capacity - constant work rate cycling test | Baseline
  Performed at 75% of maximum achieved power during two legged maximal incremental cycle test. Participants will be asked to cycle at a constant power output until volitional exhaustion. Outcome will be time (mins)
Functional capacity - measured by Timed up-and-go test | Baseline
  Time (secs) taken to get up from a chair, walk 3m, return to the chair and sit down.
Muscle strength - maximal concentric quadriceps strength | Baseline
  Isokinetic knee flexion/extension using dynamometry. Peak torque (Nm) and angle of peak torque recorded
Muscle strength - maximal eccentric quadriceps strength | Baseline
  Isokinetic knee flexion/extension using dynamometry. Peak torque (Nm) and angle of peak torque recorded
Muscle strength - 10 rep max Leg extension | Baseline
  Maximum load that participants can lift with two legs for 10 repetitions (kg)
Health related quality of life - St George's respiratory questionnaire | Baseline
  50 item questionnaire to measure health status (quality of life) in patients with diseases of airways obstruction. Scores are calculated for three domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score (from 0-100). The minimum change score of 4 units is established as clinically relevant.
Frailty - Groningen Frailty Index | Baseline
  total score out of 15. A score of 4 of more indicates moderate to severe frailty
Balance - Activities specific balance scale (ABC scale) | Baseline
  16 item score (each point answered from 0-10 with 0 representing no confidence and 100 representing complete confidence with performing specified activity without loosing balance). Total score given as an average of all questions (presented as a percentage from 0-100%). Lower scores represent worse balance
Physical activity - 7-day activity monitor | Baseline
  Percentage of time in light and moderate-to-vigorous physical activity
Muscle architectural measures seen on muscle biopsy | Baseline
  Fibre type composition - percentage of type 1 and type 2 muscle fibres
Muscle architectural measures seen on muscle biopsy | Baseline
  Fibre size - mean fibre cross sectional area (micrometer2)
Capillary density on muscle biopsy | Baseline
  Number of capillaries per mm2
Body composition - bioelectrical impedance | Baseline
  fat free mass index (kg/m2)
Breathlessness during exercise - Multidimensional dyspnoea profile | Baseline
  Validated questionnaire exploring multiple aspects of dyspnoea. Recorded at baseline and during each of 4 exercise modalities (eccentric cycling, concentric cycling, single leg cycling and lower limb resistance training). Pooled results of each question will be presented. This is not a traditional 'scale' with a 'total score' but produces a multidimensional picture of breathlessness and has been well described in breathlessness research. It is being used as a way to categorise breathlessness response or phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maltais F, Decramer M, Casaburi R, Barreiro E, Burelle Y, Debigare R, Dekhuijzen PN, Franssen F, Gayan-Ramirez G, Gea J, Gosker HR, Gosselink R, Hayot M, Hussain SN, Janssens W, Polkey MI, Roca J, Saey D, Schols AM, Spruit MA, Steiner M, Taivassalo T, Troosters T, Vogiatzis I, Wagner PD; ATS/ERS Ad Hoc Committee on Limb Muscle Dysfunction in COPD. An official American Thoracic Society/European Respiratory Society statement: update on limb muscle dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 May 1;189(9):e15-62. doi: 10.1164/rccm.201402-0373ST. PMID 24787074
- [Background] Troosters T, Gosselink R, Decramer M. Exercise training in COPD: how to distinguish responders from nonresponders. J Cardiopulm Rehabil. 2001 Jan-Feb;21(1):10-7. doi: 10.1097/00008483-200101000-00004. PMID 11271652
- [Background] Camillo CA, Osadnik CR, van Remoortel H, Burtin C, Janssens W, Troosters T. Effect of "add-on" interventions on exercise training in individuals with COPD: a systematic review. ERJ Open Res. 2016 Mar 29;2(1):00078-2015. doi: 10.1183/23120541.00078-2015. eCollection 2016 Jan. PMID 27730178
- [Background] Rocha Vieira DS, Baril J, Richard R, Perrault H, Bourbeau J, Taivassalo T. Eccentric cycle exercise in severe COPD: feasibility of application. COPD. 2011 Aug;8(4):270-4. doi: 10.3109/15412555.2011.579926. Epub 2011 Jul 5. PMID 21728805
- [Background] Bjorgen S, Helgerud J, Husby V, Steinshamn S, Richadson RR, Hoff J. Aerobic high intensity one-legged interval cycling improves peak oxygen uptake in chronic obstructive pulmonary disease patients; no additional effect from hyperoxia. Int J Sports Med. 2009 Dec;30(12):872-8. doi: 10.1055/s-0029-1238292. PMID 19821224
- [Background] Evans RA, Dolmage TE, Mangovski-Alzamora S, Romano J, O'Brien L, Brooks D, Goldstein RS. One-Legged Cycle Training for Chronic Obstructive Pulmonary Disease. A Pragmatic Study of Implementation to Pulmonary Rehabilitation. Ann Am Thorac Soc. 2015 Oct;12(10):1490-7. doi: 10.1513/AnnalsATS.201504-231OC. PMID 26291542

DOCUMENTS (1):
  • Informed Consent Form (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03817294/ICF_000.pdf